CLINICAL TRIAL: NCT07215962
Title: Real-World Long-Term Safety Outcomes and First-Line Treatment Patterns in Patients With Non-Small Cell Lung Cancer and Pd-L1 <1% in the Florida Cancer Specialists & Research Institute Database
Brief Title: Long-Term Safety Outcomes and First-Line Treatment Patterns in Patients With Non-Small Cell Lung Cancer and Programmed Death-1 (Pd-L1) <1%
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1542
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; Platinum Compounds; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Participants receiving nivolumab + ipilimumab treatment
  Interventions: Biological: Nivolumab + ipilimumab
- Cohort 2: Participants receiving nivolumab + ipilimumab + platinum-based chemotherapy
  Interventions: Biological: Nivolumab + ipilimumab + platinum-based chemotherapy
- Cohort 3: Participants receiving immuno-oncology therapy (excl nivolumab) with chemotherapy treatment
  Interventions: Biological: Immuno-oncology-based therapy (excluding nivolumab-based regimens) with chemotherapy
- Cohort 4: Participants receiving other dual-IO with chemotherapy
  Interventions: Biological: Other dual-immuno-oncology therapy with chemotherapy

INTERVENTIONS:
Biological: Nivolumab + ipilimumab — According to the product label
  Groups: Cohort 1
Biological: Nivolumab + ipilimumab + platinum-based chemotherapy — According to the product label
  Groups: Cohort 2
Biological: Immuno-oncology-based therapy (excluding nivolumab-based regimens) with chemotherapy — According to the product label
  Groups: Cohort 3
Biological: Other dual-immuno-oncology therapy with chemotherapy — According to the product label
  Groups: Cohort 4

SUMMARY:
The purpose of this study is to assess the treatment-related adverse events and associated healthcare resource use in programmed death ligand 1 (PD-L1) negative individuals diagnosed with advanced/metastatic non-small cell lung cancer (NSCLC) who received first-line therapy

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* Are ≥ 18 years of age at the index date
* Have a confirmed diagnosis of advanced/metastatic non-small cell lung cancer (NSCLC) (stage IIIB-IV) (squamous and non-squamous)
* Have PD-L1< 1% level as reported
* Received one of the following 1L treatments:

  * Cohort 1: nivolumab + ipilimumab
  * Cohort 2: nivolumab + ipilimumab + platinum-based chemotherapy
  * Cohort 3: Immuno-oncology (IO)-based therapy (excluding nivolumab-based regimens) with chemotherapy
  * Cohort 4: Dual-IO with chemotherapy (eg. tremelimumab-actl + durvalumab + carboplatin + albumin-bound paclitaxel, tremelimumab-actl + durvalumab + [carboplatin or cisplatin] + gemcitabine, tremelimumab-actl + durvalumab + carboplatin + albumin-bound paclitaxel, tremelimumab-actl + durvalumab + [carboplatin or cisplatin] + pemetrexed)
* Have ≥ 6 months of documented post-index (follow-up) period after the index date - Participants who die within 6 months of follow-up will be included

Exclusion Criteria:

* Have positive or unknown EGFR or ALK mutation before the index date
* Have a gap of > 120 days between metastatic NSCLC diagnosis and index date
* Were included in a clinical trial for 1L therapy
* Enter a hospice within 6 months of the follow-up will be excluded
* Have other concurrent primary cancer diagnoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of programmed death ligand 1 (PD-L1) negative individuals diagnosed with advanced/metastatic non-small cell lung cancer (NSCLC) who received first-line therapy in routine clinical practice at the Florida Cancer Specialists and Research Institute
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | Baseline
Participant baseline clinical characteristics | Baseline
Time to onset of treatment-related adverse events | Up to 8 years
Number of treatment-related adverse events resolved | Up to 8 years
Number of participants receiving treatment for treatment-related adverse events by drug class | Up to 8 years
Number of participants that discontinued immune-oncology therapy due to treatment-related adverse events | Up to 8 years

SECONDARY OUTCOMES:
Healthcare Resource Utilization (HCRU) associated with treatment-related adverse event | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Florida Cancer Specialists & Research Institute, Fleming Island, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts